CLINICAL TRIAL: NCT05864690
Title: Prevalence of Anxiety Disorders, Depression and Related Factors in Vietnamese Infertile Women With Polycystic Ovarian Syndrome
Brief Title: Anxiety Disorders, Depression and Related Factors in PCOS
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 04/23/DD-BVMD
Record Dates: First submitted 2023-04-18; First posted 2023-05-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: PCOS
Keywords: infertile women; PCOS; Anxiety disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Polycystic ovary syndrome (PCOS) is a systemic neuro-endocrine-metabolic-reproductive disorder, common in women of reproductive age, affecting 21.27% of women worldwide and the rate of PCOS has been increasing over the past decade.

Women with PCOS have many health problems, including insulin resistance, hyperandrogenemia, and ovulation disorders. Moreover, PCOS is also associated with significant consequences such as increased risk of cardiovascular disease, glucose intolerance and diabetes mellitus (both type 2 and gestational), increased risk of endometrial hyperplasia and endometrial cancer and mental health disorders.

A meta-analysis of 57 studies has been reported that women with PCOS are more likely to have an increased risk of diagnosis of depression, anxiety, bipolar disorder, and obsessive-compulsive disorder.

These psychological disorders may be related to biometric and biochemical characteristics in women with PCOS, such as body image, hirsutism or acne. Furthermore, researches showed that waist-to-hip ratio and plasmatic levels of testosterone is inversely related to anxiety, psychoticism, hostility and to the indexes of psychological distress. Psychological consequences may also be related to other factors, including stigmatization and isolation, the lack of empathy from family and friends, the feeling of guilt and the diminished sense of self-worth, the costs of treatment and treatment outcomes.

However, there has been no data on the psychological disorders in infertile women with PCOS. Therefore, the study aimed to determine the prevalence of anxiety disorders, depression in infertile women with PCOS and associated factors.

DETAILED DESCRIPTION:
* This trial will be conducted at My Duc Hospital, Ho Chi Minh City, Viet Nam.
* Women who are potentially eligible will be provided information about the study purposes, procedures, related risk and benefits
* Screening for eligibility will be performed on the day of the first visit when diagnosis about PCOS is established.
* Patients will be provided information related to the study together with the informed consent documents. Signed informed consent forms will be obtained by the investigators from all women before the enrolment.
* All patients selected for this study will answer the questionares and complete the GAD-7 GAD-7 (General Anxiety Disorder-7) and PHQ-9 (Patient Health Questionnaire-9) following careful instruction on how to complete the instrument by investigator in a private room without the presence of their husband.
* The survey will last about 15 minutes. If the result of the GAD-7 and PHQ-9 suggested anxiety disorders, depression, the patient will refer to specialists for further assessment and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infertile Vietnamese women
* Reporting PCOS according to Rotterdam 2003
* Agreement to participate in the study

Exclusion Criteria:

* Having a family history of neuropsychiatric disease
* Patients who are deaf, blind, or born dumb
* Patents cannot understand Vietnamese

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Infertile Vietnamese women with PCOS
Sampling Method: Non-Probability Sample
Enrollment: 768 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
The prevalence of anxiety disorders | immediately after the interview
  The prevalence of anxiety disorders using General Anxiety Disorder-7 (GAD-7). The minimum values is 0 and maximum values is 21. Using cutoff score 10 with sensitivity 89% and specificity 82% for any anxiety disorder. Higher GAD-7 scores correlate with disability and functional impairment (in measures such as work productivity and health care utilization.
The prevalence of depression | immediately after the interview
  The prevalence of depression using Patient Health Questionnaire -9 (PHQ-9). The minimum values is 0 and maximum values is 27. PHQ-9 scores ≥10 were found to be 88% sensitive and also 88% specific for detecting major depressive disorder. Higher PHQ-9 scores are associated with decreased functional status and increased symptom-related difficulties, sick days, and healthcare utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, PhD, MD, Principal Investigator — IVFMD and HOPE Research Center, My Duc Hospital
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Deswal R, Narwal V, Dang A, Pundir CS. The Prevalence of Polycystic Ovary Syndrome: A Brief Systematic Review. J Hum Reprod Sci. 2020 Oct-Dec;13(4):261-271. doi: 10.4103/jhrs.JHRS_95_18. Epub 2020 Dec 28. PMID 33627974
- [Background] Anagnostis P, Tarlatzis BC, Kauffman RP. Polycystic ovarian syndrome (PCOS): Long-term metabolic consequences. Metabolism. 2018 Sep;86:33-43. doi: 10.1016/j.metabol.2017.09.016. Epub 2017 Oct 10. PMID 29024702
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Hum Reprod. 2018 Sep 1;33(9):1602-1618. doi: 10.1093/humrep/dey256. PMID 30052961
- [Background] Brutocao C, Zaiem F, Alsawas M, Morrow AS, Murad MH, Javed A. Psychiatric disorders in women with polycystic ovary syndrome: a systematic review and meta-analysis. Endocrine. 2018 Nov;62(2):318-325. doi: 10.1007/s12020-018-1692-3. Epub 2018 Jul 31. PMID 30066285
- [Background] Borghi L, Leone D, Vegni E, Galiano V, Lepadatu C, Sulpizio P, Garzia E. Psychological distress, anger and quality of life in polycystic ovary syndrome: associations with biochemical, phenotypical andsocio-demographic factors. J Psychosom Obstet Gynaecol. 2018 Jun;39(2):128-137. doi: 10.1080/0167482X.2017.1311319. Epub 2017 Apr 6. PMID 28385114
- [Background] Authier M, Normand C, Jego M, Gaborit B, Boubli L, Courbiere B. Qualitative study of self-reported experiences of infertile women with polycystic ovary syndrome through on-line discussion forums. Ann Endocrinol (Paris). 2020 Oct;81(5):487-492. doi: 10.1016/j.ando.2020.07.1110. Epub 2020 Aug 19. PMID 32827451